CLINICAL TRIAL: NCT06496490
Title: A Phase 2 Clinical Trial of TQB2102 for Injection in Locally Advanced or Metastatic Non-small Cell Lung Cancer With HER2 Gene Abnormality to Evaluate the Efficacy and Safety
Brief Title: A Clinical Trial of TQB2102 for Injection in Non-small Cell Lung Cancer With HER2 Gene Abnormality
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-II-03
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2102 for injection (Experimental): Intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle.
  Interventions: Drug: TQB2102 for injection
- TQB2102 for injection+Benmelstobart injection (Experimental): TQB2102 for injection, intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle; Benmelstobart injection, intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle.
  Interventions: Drug: TQB2102 for injection combined with Benmelstobart injection

INTERVENTIONS:
Drug: TQB2102 for injection — HER2 dual-antibody-drug Conjugate (ADC).
  Arms: TQB2102 for injection
Drug: TQB2102 for injection combined with Benmelstobart injection — TQB2102 for injection is a HER2 dual-antibody-drug Conjugate (ADC); Benmelstobart injection is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1).
  Arms: TQB2102 for injection+Benmelstobart injection

SUMMARY:
TQB2102 is an antibody-drug conjugate comprised of a humanised antibody against Human Epidermal Growth Factor Receptor 2 (HER2), a enzyme-cleavable linker, and a topoisomerase I inhibitor payload, which combine the ability of antibodies to specifically target tumour cells with the highly potent killing activity of drugs with payloads too toxic for systemic administration. This is a Phase 2 study to evaluate the efficacy,and safety of TQB2102 for injection in locally advanced or metastatic non-small cell lung cancer with HER2 gene abnormality.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent;
* Between the ages of 18-75 years (subject to the date of signing the informed consent); Eastern cooperative oncology group (ECOG) score 0-1; estimated survival time ≥3 months;
* Patients with locally advanced, metastatic, or recurrent non-small cell lung cancer that is cytologically or histologically proven to be inoperable and cannot be treated with radical concurrent chemoradiotherapy;
* Previous standard treatments failed；
* At least one measurable lesion (based on Response Evaluation Criteria In Solid Tumors 1.1);
* Female participants of childbearing age should agree to use contraception during the study period and for 6 months after the end of the study; Have a negative serum pregnancy test within 7 days prior to study enrollment and must be a non-lactating subject; Male participants should agree that contraception must be used during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Has diagnosed and/or treated additional malignancy within 3 years prior to take medication;
* Adverse effects due to any prior treatment have not been restored to CommonTerminology Criteria for Adverse Events (CTCAE) 5.0 ≤ level 1 (Excluding hair loss);
* Major surgical treatment, incision biopsy, or significant traumatic injury were received within 28 days prior to study treatment,and minor traumatic surgery (biopsy, bronchoscopy, and chest drainage) within 7 days;
* Long-term unhealed wounds or fractures;
* History of interstitial lung disease, radiation pneumonia, and immune-related pneumonia treated with steroids in the past, or active non-infectious pneumonia with interstitial changes such as interstitial lung disease, radiation pneumonia, and immune-related pneumonia in the screening period, active pulmonary tuberculosis, pneumoconiosis, or other types of pneumonia ≥ grade 2, or severe impairment of lung function confirmed by pulmonary function examination;
* Arterial/deep vein thrombosis events occurred within 6 months prior to treatment, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism;
* Patients who have a history of psychotropic substance abuse and are unable to abstain or have mental disorders;
* Patients with any severe and/or uncontrolled disease;
* Any anticancer therapy or any other investigational drug treatment within 28 days or 5 half-lives prior to the first dosing of this study;
* Within 1 week prior to the first administration of this study, the Chinese patent drugs with anti-tumor indications clearly stated in the National MedicalProducts Administration approved drug instructions were treated;
* Local focal palliative radiotherapy was received within 2 weeks before the first dose;
* Patients with serous effusion requiring repeated drainage to relieve clinical symptoms or who have received serous effusion drainage for therapeutic purposes within 2 weeks prior to treatment;
* There is symptomatic or progressive exacerbation of central nervous system metastatic or cancerous meningitis with diffuse spread. Subjects with a history of brain metastases may be considered for inclusion if they are clinically stable;
* Severe bone injury caused by tumor bone metastasis, including pathological fractures and spinal cord compression that occurred within 6 months or are likely to occur in the near future;
* Pain associated with uncontrolled bone metastases;
* Allergic to humanized monoclonal antibody products;
* Allergic to any investigational drug or to any ingredient or excipient in the drug;
* Persons who have received live attenuated vaccine within 4 weeks prior to treatment;
* Subjects who, in the investigator's judgment, have concomitant diseases that seriously endanger the safety of subjects or interfere with the completion of the study, or who are deemed unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to 8 months
  ORR defined as percentage of participants achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Duration Of Remission (DOR) | Baseline up to 8 months
  DOR defined as the time when the participants first achieved complete or partial remission to disease progression.
Progression-Free Survival (PFS) | Baseline up to 8 months
  PFS defined as the time from the first injection until the first documented progressive disease (PD) or death from any cause, whichever happens first.
Overall Survival (OS) | Baseline up to 18 months
  OS defined as the time from the first injection to death from any cause.
Frequency of adverse event (AE) | From the date of signing the informed consent to 28 days after the last dosing or a new anti-tumor treatment, whichever comes first.
  The occurrence of all adverse medical events after the first injection.
Severity of adverse event (AE) | From the date of signing the informed consent to 28 days after the last dosing or a new anti-tumor treatment, whichever comes first.
  The severity of all adverse medical events after the first injection.
Anti-drug antibody (ADA) | Before infusion on Cycle1 Day1, Cycle2 Day1, Cycle 4 Day1, Cycle7 Day1, Cycle12 Day1 (each cycle is 21 days), 90 days after the end of the last infusion (each cycle is 21 days).
  Incidence of anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Foshan First People's Hospital, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The Second Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Harbin Medical University cancer hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Provincial Tumor Hospital, Changsha, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Leshan People's Hospital, Leshan, Sichuan
  - Xinjiang Uygur Autonomous Region Cancer Hospital, Ürümqi, Xinjiang
  - The 1th School of Medicine,School of Information and Engineering.The 1th Affiliated Hospital of WMU, Wenzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University Cancer Institute&Hpspital, Tianjin